CLINICAL TRIAL: NCT00881049
Title: Phase II Trial of Imatinib(Gleevec®) in Selected Patients With Metastatic Melanoma
Brief Title: Trial of Imatinib (Gleevec®) in Selected Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Jun Guo, Beijing Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571BCN19T
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2011-01

CONDITIONS: Metastatic Melanoma
Keywords: metastatic acral or mucosal melanoma with c-kit mutation or copy number increase
MeSH Terms: conditions — Melanoma | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Imatinib (Gleevec) — Imatinib will be given for enrolled patients to investigate efficacy and safety

SUMMARY:
This study is a single-armed, open-label, single-center phase II trial of signal transduction inhibitor number 571 (STI-571) systemic therapy in selective patients with metastatic melanoma, and aims to study the efficacy and safety. The primary endpoint is progression-free survival (PFS) and the second endpoints are overall response rate (ORR), overall survival (OS), 1-year OS and safety.

DETAILED DESCRIPTION:
Only patients who meet the inclusion and exclusion criteria will be enrolled. The estimated recruitment duration is 1 year. Imatinib will be given in the dose of 400 mg orally each day unless disease progression or intolerance. The follow-up is 12 months.

Forty-eight subjects will be recruited for this study. This sample size is justified by the number of patients required to establish an improvement in PFS with statistical significance compared to historical control.

The standardized RECIST (Response Evaluation Criteria in Solid Tumors) method of unidimensional tumor assessment will be employed to evaluate tumor lesion size per 2 months in the determination of response rate and progression free survival. Repeated radiographic assessment at 4 week intervals is consistent with general oncological practice associated with computerized tomography (CT) or magnetic resonance imaging (MRI) scan testing. All efficacy endpoints will be evaluated by the investigator.

Safety will be characterized in terms of the incidence, timing, severity, and relatedness of adverse events and laboratory abnormalities. Severity will be graded according to the NCI CTCAE Version 3.0.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed melanoma with metastases and has no received any systemic treatment within 1 month
2. Evidence of mutations and/or copy number increases of KIT with laboratory examination documented from either primary or metastatic tumor site
3. ECOG performance status 0, 1, or 2
4. Estimated life expectancy of 6 months or greater
5. Age 18 years or older, male of female
6. At least one measurable site of disease
7. Adequate organ function
8. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

1. Melanoma from primary sites other than acral or mucosal melanoma
2. Received systemic anti-cancer therapy within 1 month before enrollment for metastatic disease
3. Diagnosis of any second malignancy within the last 5 years, except for adequately treated basal cell carcinoma, squamous cell skin cancer, or in situ cervical cancer
4. Severe and/or uncontrolled concomitant medical diseases
5. pregnant or childbreeding women
6. Known hypersensitivity to imatinib
7. Current treatment on another clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2008-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Bejing, China